CLINICAL TRIAL: NCT05423340
Title: A Randomized, Parallel-group Open-label Trial of ENDS Users Switching From Flavors of Potentially High-toxicity Profile to Flavors of Potentially Low-toxicity Profile (CRoFT_3.2)
Brief Title: Effect of E-Liquid Flavor on Respiratory Symptoms in People Using Electronic Nicotine Delivery Systems
Acronym: CRoFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: University of Rochester (Other); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I 2588022; U54CA228110 (NIH)
Record Dates: First submitted 2022-06-03; First posted 2022-06-21 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Electronic Cigarette Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Use Own Brand of Flavored Product (Experimental): Participants will use their current flavor of e cigarettes for 90 days
  Interventions: Other: E-cigarette Flavor
- Use Provided Tobacco Flavor (Experimental): Participants will use a new assigned flavor for 90 days
  Interventions: Other: E-cigarette Flavor
- Vaping Abstinence - use "Tobacco Free" Nicotine Pouches (Active Comparator): Participants will be asked to stop vaping for 90 days and instead only use the provided 'tobacco free' nicotine pouches.
  Interventions: Other: Tobacco Free Nicotine Pouch

INTERVENTIONS:
Other: E-cigarette Flavor — Participants use an electronic nicotine delivery system with an assigned tobacco-flavored e-liquid
  Arms: Use Own Brand of Flavored Product; Use Provided Tobacco Flavor
Other: Tobacco Free Nicotine Pouch — participants will use tobacco free oral nicotine pouches
  Arms: Vaping Abstinence - use "Tobacco Free" Nicotine Pouches

SUMMARY:
This is a randomized, parallel-group open-label trial to evaluate respiratory symptoms in ENDS users switching from banned flavors to a non-banned flavor (tobacco) or 'tobacco free' nicotine pouches.

ELIGIBILITY:
Inclusion Criteria:

* ENDS users as determined by: (a) using banned flavored ENDS with nicotine such as fruit, candy, dessert flavors, and/or any product that indicates such flavors (b) using ENDS daily, regularly for the past 6 months (self-reported).
* No smoking tobacco or using smokeless tobacco for the past 6 months.
* Subjects should be free of acute respiratory illness within the proceeding 30 days prior to recruitment (self-reported).
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.
* After receiving information regarding the NYS flavor ban individuals must not want to quit vaping or stop using their flavored product for the next 90 days.

Exclusion Criteria:

* Individuals with health conditions and therapies that may affect immune responses and levels of inflammatory markers, including allergic rhinitis, aspirin/NSAID therapy, asthma, immunodeficiency (HIV or other), Guillain-Barre Syndrome, COPD, or fever/respiratory illness within 30 days prior to entry into study (self-reported).
* Pregnant or nursing female participants (self-reported on telephone screener, pregnancy test on Visit#1)
* Unable to communicate in English.
* Unable or unwilling to follow protocol requirements.
* Self-report having active, untreated medical/psychiatric conditions.
* History of serious side effects from nicotine or from any nicotine replacement therapies.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Vulnerable populations, such as cognitively impaired adults, individuals who are not yet adults, pregnant women, and prisoners.
* Any condition which in the Investigator's opinion deems the participant an unsuitable candidate to receive study drug.
* After receiving information about the NYS flavor ban, participants who report that they are thinking about quitting or stop using their flavor within the next 90 days.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 163 (Actual)
Dates: Start 2022-06-12 (Actual); Primary Completion 2024-10-03 (Actual); Study Completion 2024-10-03 (Actual)

PRIMARY OUTCOMES:
Risk biomarkers of inflammation and oxidative stress as measured by ELISA | Up to 90 days
  Oxidative stress and inflammation in plasma using ELISA . A quantitative measure of expression (units:pg/mg) will be produced.
Respiratory tract inflammation activity | Up to 90 days
  Exhaled Nitric Oxide (FeNo)l be measured in participants' breath using a FDA cleared monitor NIOX VERO (Aerocrine) according to ATS guidelines. FeNO has been used to monitor airway inflammation to account for persistent and/or high allergen exposure as a factor associated with higher levels of FeNO

SECONDARY OUTCOMES:
Amount of recent flavored product use | UP to 90 days
  Assessed using the PhenX Toolkit which tracks tobacco use and asks subjects to retrospectively estimate product use,
Flavor Preference questionnaire | Up to 90 days
  Personal flavor questionnaire to determine flavor preference when using ENDS.
Frequency of flavored product use | Up to 90 days
  Questions from Wave 1 Adult PATH Survey to measure use and regularity of use flavored products

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Goniewicz, PhD, Principal Investigator — Roswell Park
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT05423340/ICF_000.pdf